CLINICAL TRIAL: NCT00090779
Title: The SETPOINT Study - A Randomized Study of the Effect of Immediate Treatment With Potent Antiretroviral Therapy Versus Observation With Treatment as Indicated in Newly Infected HIV-1 Infected Subjects: Does Early Therapy After the Virologic Setpoint?
Brief Title: Nine Month Course of Anti-HIV Medications for People Recently Infected With HIV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The DSMB concluded that the findings regarding the primary analysis would persist and that no additional study goals would be achieved by continuing the study.
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Adult AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5217; 1U01AI068636 (NIH); AIEDRP AIN503; ACTG A5217
Record Dates: First submitted 2004-09-03; First posted 2004-09-06 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IT arm (Active Comparator): IT (immediate treatment) arm participants received emtricitabine/tenofovir disoproxil fumarate once daily and lopinavir/ritonavir twice daily
  Interventions: Drug: Emtricitabine/ tenofovir disoproxil fumarate; Drug: Lopinavir/Ritonavir
- DT arm (No Intervention): DT (deferred treatment) arm participants received no treatment

INTERVENTIONS:
Drug: Emtricitabine/ tenofovir disoproxil fumarate — once daily
  Arms: IT arm
Drug: Lopinavir/Ritonavir — twice daily
  Arms: IT arm

SUMMARY:
Although some doctors favor starting anti-HIV treatment as soon as possible after patients learn they are infected, it is not known if treatment for recently infected patients results in long-term benefits or harm. The purpose of this study is to learn whether or not people should take anti-HIV drugs when they are first infected.

DETAILED DESCRIPTION:
Combination antiretroviral therapy has resulted in significantly decreased morbidity and mortality, incidence of opportunistic infections, and hospitalizations in HIV infected people. However, because of long-term toxicities associated with long-term use of antiretrovirals and the persistence of virus in latent reservoirs, it is unclear when it is best to initiate therapy in recently infected individuals. This study compared the virologic outcomes of adults recently infected with HIV who received emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), coformulated as Truvada, and lopinavir/ritonavir (LPV/RTV), coformulated as Kaletra [immediate treatment (IT arm)], with those who received no treatment [deferred treatment (DT arm)].

The original study lasted 96 weeks. Participants were randomly assigned to one of two groups (IT arm vs. DT arm). For the first 36 weeks of the study, IT arm participants received FTC/TDF once daily and LPV/RTV twice daily. Some IT arm participants received a different ART regimen as determined by the participant and study staff, if appropriate. DT arm participants received no treatment for the duration of the study. At Week 37, participants from both arms were offered treatment continuation or initiation until Week 96 if they had a high viral load, low CD4 count, or experienced HIV-related symptoms (Step 2). Study visits occurred at screening, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 37, 38, 40, and every 4 weeks thereafter. Clinical assessment and blood collection occurred at all visits. Urine tests occurred at selected visits. Participants were asked to complete an adherence questionnaire at Weeks 12, 24, and 36.

Per the recommendations the DSMB review in June 2009, this protocol was terminated as originally written with the exception of those participants in the IT arm in the middle of the first 36 weeks of treatment. Those participants were to continue on treatment until the end of the 36 weeks. At that point treatment decisions were made on best practice guidelines. In addition, the study duration was extended to include a 5 year follow up of participants who did not initiate long-term antiretroviral therapy (Step 3).

The study was reviewed by an SMC on December 8, 2010. The SMC recommended the study close to long term follow-up because only very few participants enrolled in this portion of the study.

All the results except for the CD4 analysis and time to treatment initiation and deaths were based on the database frozen on July 2, 2009. The results for the CD4 analysis and time to treatment initiation and deaths were based on the database frozen on January 30, 2012.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* Recently infected with HIV
* No prior antiretroviral therapy (ART)
* CD4 count of 350 cells/mm3 or more AND a CD4% of 14% or more within 21 days prior to study entry
* HIV viral load of 500 copies/ml or more within 21 days prior to study entry
* Required laboratory values obtained within 21 days prior to study entry
* 18 years or older
* Ability and willingness to provide written informed consent
* Willing to use acceptable forms of contraception

Exclusion Criteria for Step 1:

* HIV progression to CDC category B or C disease
* Pregnancy or breastfeeding
* History of pancreatitis or coronary artery disease
* Prior ART. Participants who took antiretrovirals for postexposure prophylaxis more than one year prior to study entry are not excluded.
* Certain medications within 21 days prior to study entry. Participants who agree to receive an alternative ART regimen approved by the investigator will not be excluded.
* Previously received an investigational anti-HIV vaccine
* Current therapy with systemic corticosteroids. Patients who are taking a short course (less than 21 days) of corticosteroids are not excluded.
* Current therapy with systemic chemotherapeutic agents; nephrotoxic systemic agents; immunomodulatory treatments, including interleukin-2; or investigational agents
* Known allergy or sensitivity to study drugs or their formulations
* Current alcohol or drug use that, in the opinion of the investigator, would interfere with the study
* Serious medical or psychiatric illness that, in the opinion of the investigator, would interfere with the study
* Hepatitis B surface antigen positive within 21 days prior to study entry
* Known resistance to one or more components of the study drug regimen

Inclusion Criteria for Step 2:

* subjects in DT arm who meet one of the following five criteria will be advised to enter step 2 and initiate ART:

  1. CD4 cell counts below 350 cells/mm3 on 2 consecutive determinations at least 4 weeks apart at or after the step 1, week 12 study visit
  2. HIV-1 RNA above 750,000 copies/mL confirmed on 2 consecutive determinations at least 1 week apart at or after the step 1, week 4 study visit
  3. HIV-1 RNA above 200,000 copies/mL on 2 consecutive determinations at least 1 week apart at or after the step 1, week 12 study visit
  4. Clinical progression to CDC category B or C disease
  5. CD4 count below 200 cells/mm3 or CD4 percent less than 14% at any time on study
* subjects in IT arm who meet one of the following five criteria after discontinuing study medications will be advised to enter step 2 and re-initiate ART:

  1. CD4 cell counts below 350 cells/mm3 on 2 consecutive determinations at least 4 weeks apart at or after the step 1, week 12 post-treatment- discontinuation study visit
  2. HIV-1 RNA above 750,000 copies/mL confirmed on 2 consecutive determinations at least 1 week apart at or after the step 1, week 4 post-treatment- discontinuation study visit
  3. HIV-1 RNA above 200,000 copies/mL on 2 consecutive determinations at least 1 week apart at or after the step 1, week 12 post-treatment- discontinuation study visit
  4. Clinical progression to CDC category B or C disease
  5. CD4 count below 200 cells/mm3 or CD4 percent less than 14% at any time on study

     Exclusion Criteria for Step 2:
* Pregnancy or breastfeeding

Inclusion Criteria for Step 3:

* Study participants who were on Step 1, IT arm and had completed or ended prematurely the 36 week course of early ART and did not on ART either because they did not meet eligibility criteria for Step 2 or because they did not start ART even after meeting the Step 2 eligibility criteria.
* Study participants on Step 1, DT arm who were not on ART either because they did not meet eligibility criteria for Step 2 or because they did not start ART even after meeting the Step 2 eligibility criteria.
* Previous A5217 participants who had either completed the study or ended prematurely their participation in the study, AND were not on ART either because they never met eligibility criteria for Step 2 or because they had not started ART even after meeting the Step 2 eligibility criteria.
* All A5217 participants who were on Step 1 and in the midst of their 36 weeks of randomized ART and who completed a portion or all of the 36 weeks of originally recommended therapy, AND chose then to interrupt their ART.

Exclusion Criteria for Step 3:

* Participants who were on Step 1, IT arm of the study receiving ART.
* Participants in Step 2 or who had otherwise initiated long-term ART, regardless of whether they were on treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-01; Primary Completion 2009-07 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hogan, MD, Study Chair — Division of Infectious Diseases, Columbia University College of Physicians and Surgeons
Locations (27):
- United States (25):
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - University of Miami AIDS CRS (901), Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Indiana University Hospital (2601), Indianapolis, Indiana
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - HIV Prevention & Treatment CRS (30329), New York, New York
  - AIDS Care CRS (1108), Rochester, New York
  - University of Rochester ACTG CRS (1101), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Moses H. Cone Memorial Hospital CRS (3203), Greensboro, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS (3203), Greensboro, North Carolina
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
  - University of Washington AIDS CRS (1401), Seattle, Washington
  - UW Primary Infection Clinic CRS (1404), Seattle, Washington
- Peru (2):
  - San Miguel CRS, San Miguel, Lima region
  - Asociacion Civil Impacta Salud y Educacion - Miraf CRS (11301), Lima

REFERENCES:
- [Background] Fidler S, Oxenius A, Brady M, Clarke J, Cropley I, Babiker A, Zhang HT, Price D, Phillips R, Weber J. Virological and immunological effects of short-course antiretroviral therapy in primary HIV infection. AIDS. 2002 Oct 18;16(15):2049-54. doi: 10.1097/00002030-200210180-00010. PMID 12370504
- [Background] Kassutto S, Rosenberg ES. Primary HIV type 1 infection. Clin Infect Dis. 2004 May 15;38(10):1447-53. doi: 10.1086/420745. Epub 2004 Apr 30. PMID 15156484
- [Background] Little SJ, Holte S, Routy JP, Daar ES, Markowitz M, Collier AC, Koup RA, Mellors JW, Connick E, Conway B, Kilby M, Wang L, Whitcomb JM, Hellmann NS, Richman DD. Antiretroviral-drug resistance among patients recently infected with HIV. N Engl J Med. 2002 Aug 8;347(6):385-94. doi: 10.1056/NEJMoa013552. PMID 12167680
- [Background] Pilcher CD, Eron JJ Jr, Galvin S, Gay C, Cohen MS. Acute HIV revisited: new opportunities for treatment and prevention. J Clin Invest. 2004 Apr;113(7):937-45. doi: 10.1172/JCI21540. PMID 15057296
- [Result] Messer K, Vaida F, Hogan C. Robust analysis of biomarker data with informative missingness using a two-stage hypothesis test in an HIV treatment interruption trial: AIEDRP AIN503/ACTG A5217. Contemp Clin Trials. 2006 Dec;27(6):506-17. doi: 10.1016/j.cct.2006.07.003. Epub 2006 Jul 25. PMID 16962381
- [Result] Hogan CM, Degruttola V, Sun X, Fiscus SA, Del Rio C, Hare CB, Markowitz M, Connick E, Macatangay B, Tashima KT, Kallungal B, Camp R, Morton T, Daar ES, Little S; A5217 Study Team. The setpoint study (ACTG A5217): effect of immediate versus deferred antiretroviral therapy on virologic set point in recently HIV-1-infected individuals. J Infect Dis. 2012 Jan 1;205(1):87-96. doi: 10.1093/infdis/jir699. Epub 2011 Dec 15. PMID 22180621
- See also: Click here for more information about the AIEDRP CORE01 study — http://clinicaltrials.gov/ct/show/NCT00086372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 27 study sites (25 in the US and 2 in Peru) in the AIDS Clinical Trials Group system between February 2005 and June 2009.
Groups:
- IT Arm: On step 1, IT arm participants received 36 weeks of emtricitabine/tenofovir disoproxil fumarate once daily and lopinavir/ritonavir twice daily. Participants in IT arm who met clinical, virologic or immunologic criteria for treatment re-initiation entered step 2 and re-initiated ART. At the time of the end of original randomized study, study participants in IT arm who did not enter Step 2 and did not initiate ART without meeting eligibility criteria for Step 2 had the opportunity to take part in a long-term follow-up study (step 3) for up to a total duration of five years in order to ascertain information about HIV-1 RNA, CD4+ T-cell count, occurrence of CDC Category B or C diagnoses, and initiation of ART.
- DT Arm: On step 1, DT arm participants received no Treatment,unless subsequent disease progression criteria were met. Participants in DT arm who met clinical, virologic or immunologic criteria for treatment initiation entered step 2 and initiated ART. At the time of the end of original randomized study, study participants in DT arm who did not enter Step 2 and did not initiate ART without meeting eligibility criteria for Step 2 had the opportunity to take part in a long-term follow-up study (step 3) for up to a total duration of five years in order to ascertain information about HIV-1 RNA, CD4+ T-cell count, occurrence of CDC Category B or C diagnoses, and initiation of ART.
Period: Step 1
Arm/Group | IT Arm | DT Arm
Started | 66 | 64
Completed | 55 (Results are based on the database frozen on July 2, 2009 per DSMB recommendation of study closure.) | 49 (Results are based on the database frozen on July 2, 2009 per DSMB recommendation of study closure.)
Not Completed | 11 | 15
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Non-compliance to study requirements | 0 | 1
Not completed — Subject relocated | 2 | 8
Period: Step 2
Arm/Group | IT Arm | DT Arm
Started | 6 (One subject who had two consecutive CD4<350cells/mm^3 did not enter step 2.) | 19 (Three with two consecutive CD4<350cells/mm^3 and one with CDC category B event didn't enter step 2.)
Completed | 0 | 1
Not Completed | 6 | 18
Not completed — Off study per study closure | 6 | 16
Not completed — Subject relocated | 0 | 1
Not completed — Non-compliance to study requirements | 0 | 1
Period: Step 3
Arm/Group | IT Arm | DT Arm
Started | 7 | 5
Completed | 0 | 0
Not Completed | 7 | 5
Not completed — Initiation of ART and off extended study | 3 | 2
Not completed — Off extended study due to study closure | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- IT Arm: IT arm participants received emtricitabine/tenofovir disoproxil fumarate once daily and lopinavir/ritonavir twice daily
- DT Arm: DT arm participants received no Treatment
- Total: Total of all reporting groups
Arm/Group | IT Arm | DT Arm | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (11.3) | 34.6 (9.1) | 34.4 (10.3)
Age, Customized [Number; unit: participants]
  <20 years | 4 | 0 | 4
  20-29 years | 24 | 23 | 47
  30-39 years | 19 | 21 | 40
  40-49 years | 12 | 16 | 28
  50-59 years | 4 | 4 | 8
  60-69 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 58 | 59 | 117
Race [Number; unit: participants]
  White | 49 | 56 | 105
  Black/ African American | 10 | 3 | 13
  Other | 4 | 4 | 8
  Unknown | 3 | 1 | 4
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 52 | 55 | 107
CD4 Counts [Mean (Standard Deviation); unit: cells/mm3] | 570 (197) | 611 (207) | 590 (202)
CD4 Count Category [Number; unit: participants]
  201-350 cells/mm^3 | 4 | 2 | 6
  351-500 cells/mm^3 | 26 | 24 | 50
  >500 cells/mm^3 | 36 | 38 | 74
Log10 HIV-1 RNA Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] | 4.4 (0.6) | 4.4 (0.6) | 4.4 (0.6)
HIV-1 RNA Viral Load Category [Number; unit: participants]
  200-399 copies/mL | 0 | 1 | 1
  400-999 copies/mL | 1 | 0 | 1
  1000-9999 copies/mL | 16 | 15 | 31
  >=10000 copies/mL | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Ranked Log10 HIV-1 RNA Viral Load (log10 Copies/mL) Averaged at 72 and 76 Weeks for the IT Arm and DT Arm
Description: The primary endpoint is (i) the average of log10 viral loads (VL) at wks 72 and 76 for participants who continued to wk 72 off ARV for the DT arm, (ii) average wk 72 and 76 VL for those who continued to wk 36 off ARV for the IT arm and (iii) an assigned VL rank for the "failures" who needed ARVs or met criteria for entry into Step 2 prior to these study visits. The assigned rank for the failures was either the last observed rank carried forward or the worst rank relative to the other possible outcomes. This approach was designed to, if anything, bias against finding a treatment effect. To illustrate, consider five participants who enter the study (A, B, C, D, and E), 4 of whom (A, B, C, D) make it to 72 wks off therapy with RNA levels that increase from A to D. Participant E enters Step 2 at wk 12, at which time his RNA is in the 50th percentile. This rank would be carried forward, so the rank order of the log10 HIV-1 RNA endpoints would be A B E C D.
Time Frame: At Weeks 72 and 76
Population: Participants in follow-up at least 72 weeks since randomization were included.
Measure: Median (Full Range); unit: rank
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 39 | 40
rank | 26.0 [1.0 to 70.0] | 49.3 [4.0 to 70.0]
Statistical Analysis 1: Comparison: IT Arm vs DT Arm; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Ranked log10 HIV-1 RNA Viral Load (log10 Copies/mL) Averaged at Weeks 72 and 76 for the IT Arm and Ranked log10 HIV-1 RNA Viral Load (log10 Copies/mL) Averaged at Weeks 36 and 40 for the DT Arm
Description: The primary endpoint is (i) average wk 36 and 40 VL for those who continued to wk 36 off ARV for the DT arm, (ii) average wk 72 and 76 VL for those who continued to wk 36 off ARV for the IT arm and (iii) an assigned VL rank for the "failures" who needed ARVs or met criteria for entry into Step 2 prior to these study visits. The assigned rank for the failures was either the last observed rank carried forward or the worst rank relative to the other possible outcomes. This approach was designed to, if anything, bias against finding a treatment effect. To illustrate, consider five participants who enter the study (A, B, C, D, and E), 4 of whom (A, B, C, D) make it to 72 wks off therapy with RNA levels that increase from A to D. Participant E enters Step 2 at wk 12, at which time his RNA is in the 50th percentile. This rank would be carried forward, so the rank order of the log10 HIV-1 RNA endpoints would be A B E C D.
Time Frame: IT arm (weeks 72 and 76) and DT arm ( weeks 36 and 40)
Population: Participants in follow-up at least 72 weeks since randomization were included.
Measure: Median (Full Range); unit: rank
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 39 | 40
rank | 26.0 [1.0 to 70.0] | 48.5 [28.0 to 67.5]
Statistical Analysis 1: Comparison: IT Arm vs DT Arm; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Participants Experiencing Either a CDC Category B or C Diagnosis, CD4<200 Cells/mm^3 or CD4 Percent <14%.
Time Frame: 96 weeks since randomization
Measure: Number; unit: participants
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 66 | 64
participants | 2 | 8

4. Secondary Outcome: Change in CD4 Counts Cells/mm^3 From Week 36 for IT Arm and From Week 0 for DT Arm
Time Frame: IT arm (weeks 36, 60, 72, 84 and 96) and DT arm (weeks 0, 24, 36, 48 and 60)
Population: One subject in IT arm with multidrug resistance at baseline was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Change in Log10 transformed CD4 Counts
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 65 | 64
Change in Log10 transformed CD4 Counts
  IT arm (wk 60- wk 36) vs. DT arm (wk 24- wk 0) | -0.11 (0.10) | -0.02 (0.12)
  IT arm (wk 72- wk 36) vs. DT arm (wk 36- wk 0) | -0.10 (0.12) | -0.03 (0.11)
  IT arm (wk 84- wk 36) vs. DT arm (wk 48- wk 0) | -0.10 (0.12) | -0.06 (0.17)
  IT arm (wk 96- wk 36) vs. DT arm (wk 60- wk 0) | -0.12 (0.13) | -0.02 (0.15)

5. Secondary Outcome: Number of Participants Meeting Clinical, Virologic, or Immunologic Criteria for Treatment Initiation or Re-initiation
Description: The clinical, virologic, or immunologic criteria for treatment initiation or re-initiation include CD4 count below 350 cells/mm^3 on two consecutive determinations at least 4 weeks apart, at least 12 weeks into the study or 12 weeks post-treatment discontinuation, (2) confirmed CD4 count below 200 cells/mm^3 or CD4 percent below 14% at any time on study, (3) confirmed HIV-1 RNA level above 750,000 copies/mL 4 weeks into the study or above 200,000 copies/mL 12 weeks or more into the study, or (4) CDC Category B or C diagnosis.
Time Frame: 96 weeks since randomization
Population: All 130 eligible subjects were included.
Measure: Number; unit: Participants
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 66 | 64
Participants | 7 | 23

6. Secondary Outcome: Number of Participants in IT Arm Off Treatment Before 36 Weeks
Description: The study provided fixed-dose combination emtricitabine/tenofovir DF 200/300 mg orally once daily and lopinavir/ritonavir 200/50 mg administered either as two tablets twice daily or four tablets once daily, for the first 36 weeks for individuals in the IT arm.
Time Frame: At Week 36
Population: All 66 eligible subjects in IT arm were included.
Measure: Number; unit: participants
Arm/Group | IT Arm
Number analyzed (Participants) | 66
participants | 8

7. Secondary Outcome: Time to Meeting the Clinical, Virologic, or Immunologic Criteria for Treatment Initiation or Re-initiation
Description: 5th, 10th, 25th, 50th, 75th and 90th percentiles in weeks from randomization to meeting the criteria for treatment initiation or re-initiation which include CD4 count below 350 cells/mm^3 on two consecutive measurements at least 4 weeks apart, at least 12 weeks into the study or 12 weeks post-treatment discontinuation, confirmed CD4 count below 200 cells/mm^3 or CD4 percent below 14% at any time on study, confirmed HIV-1 RNA level above 750,000 copies/mL 4 weeks into the study or above 200,000 copies/mL 12 weeks or more into the study, or CDC Category B or C diagnosis.
Time Frame: 96 weeks since randomization
Population: Throughout database cutoff for DSMB review (by July 2, 2009).
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 65 | 64
weeks
  5th percentile | 6.3 [0 to 13.0] | 6.9 [2.3 to 12.3]
  10th percentile | 13.0 [0 to 26.1] | 12.3 [2.3 to 18.3]
  25th percentile | 36.4 [19.9 to 50.4] | 26.3 [16.9 to 36.4]
  50th percentile | 72.0 [52.4 to 94.1] | 60.0 [36.4 to 93.9]
  75th percentile | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 25% | 96.0 [72.0 to 96.0]
  90th percentile | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 10% | 96.0 [96.0 to NA] — Not estimable as the upper limit for survival function at all weeks is above 10%

8. Secondary Outcome: Time From Study Entry in DT Arm Participants or From Week 36 in IT Arm Participants to Meeting the Clinical, Virologic, or Immunologic Criteria for Treatment Initiation or Re-initiation
Description: 5th, 10th, 25th, 50th, 75th and 90th percentiles in weeks from randomization for DT arm or from week 36 for IT arm to meeting the criteria for treatment initiation or re-initiation which include two consecutive CD4 count below 350 cells/mm^3 at least 4 weeks apart, at least 12 weeks into the study or 12 weeks post-treatment discontinuation, confirmed CD4 count below 200 cells/mm^3 or CD4 percent below 14% at any time on study, confirmed HIV-1 RNA level above 750,000 copies/mL 4 weeks into the study or above 200,000 copies/mL 12 weeks or more into the study, or CDC Category B or C diagnosis.
Time Frame: 96 weeks since randomization
Population: Through database cutoff for DSMB review (by July 2, 2009). The analysis includes only those in the IT arm who continued ART through week 36 (n=49), compared to all in the DT arm (n=64).
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 65 | 64
weeks
  5th percentile | 5.1 [0.4 to 13.0] | 6.9 [2.3 to 12.3]
  10th percentile | 10.4 [0.4 to 16.4] | 12.3 [2.3 to 18.3]
  25th percentile | 22.7 [13.0 to 39.3] | 26.3 [16.9 to 36.4]
  50th percentile | 58.1 [36.0 to NA] — Not estimable as the upper limit for survival function at all weeks is above 50% | 60.0 [36.4 to 93.9]
  75th percentile | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 25% | 96.0 [72.0 to 96.0]
  90th percentile | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 10% | 96.0 [96.0 to NA] — Not estimable as the upper limit for survival function at all weeks is above 10%

9. Secondary Outcome: Time to Treatment Initiation or Death
Description: 5th, 10th, 25th, 50th and 75th percentiles in weeks from randomization to treatment initiation or death
Time Frame: 5 years since randomization
Population: All eligible subjects were included except one subject in IT arm with baseline multidrug resistance.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | IT Arm | DT Arm
Number analyzed (Participants) | 65 | 64
weeks
  5th percentile | 36 [0 to 36.9] | 13.9 [6.4 to 20.9]
  10th percentile | 36.9 [0 to 51.9] | 20.9 [6.4 to 37.0]
  25th percentile | 67.1 [44.0 to 94.6] | 43.7 [31.6 to 96.0]
  50th percentile | 96.4 [94.0 to 157.9] | 97.3 [94.0 to 146.4]
  75th percentile | 163.3 [97.7 to NA] — Not estimable as the upper limit for survival function at all weeks is above 25% | 157.7 [99.9 to NA] — Not estimable as the upper limit for survival function at all weeks is above 25%

ADVERSE EVENTS:
Time Frame: 5 years since randomization
Arm/Group | IT Arm | DT Arm
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/64
Other Adverse Events (participants affected / at risk) | 58/66 | 48/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IT Arm (N=66) | DT Arm (N=64)
Blood bilirubin increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IT Arm (N=66) | DT Arm (N=64)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 19 | 10
Nausea (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 5 | 4
Fatigue (General disorders) | 9 | 6
Pyrexia (General disorders) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 4
Alanine aminotransferase increased (Investigations) | 10 | 15
Aspartate aminotransferase increased (Investigations) | 8 | 12
Blood bilirubin increased (Investigations) | 7 | 3
Blood cholesterol abnormal (Investigations) | 15 | 12
Blood cholesterol increased (Investigations) | 13 | 10
Blood glucose abnormal (Investigations) | 9 | 10
Blood glucose decreased (Investigations) | 7 | 5
Blood phosphorus decreased (Investigations) | 22 | 12
Blood triglycerides abnormal (Investigations) | 4 | 4
Blood uric acid increased (Investigations) | 5 | 2
Lipase increased (Investigations) | 6 | 13
Low density lipoprotein (Investigations) | 3 | 5
Low density lipoprotein abnormal (Investigations) | 15 | 17
Low density lipoprotein increased (Investigations) | 9 | 3
Neutrophil count decreased (Investigations) | 6 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 4 | 5
Migraine (Nervous system disorders) | 4 | 0
Depression (Psychiatric disorders) | 6 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 4
Hypertension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights".